CLINICAL TRIAL: NCT02213926
Title: An Open-label, Phase 2 Study of ACP-196 in Subjects With Mantle Cell Lymphoma
Brief Title: An Open-label, Phase 2 Study of ACP-196 (Acalabrutinib) in Subjects With Mantle Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACE-LY-004; 2023-509352-34-00 (Registry Identifier: EU CTIS); 2014-002117-28 (EudraCT Number)
Record Dates: First submitted 2014-08-05; First posted 2014-08-12 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Mantle Cell Lymphoma (MCL)
Keywords: Bruton tyrosine kinase inhibitor; Btk; Mantle Cell Lymphoma; MCL; ACP-196; Acalabrutinib; ACE-LY-004; Calquence
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ACP-196 (acalabrutinib) Regimen 1 (Experimental): ACP-196 (acalabrutinib) Regimen 1
  Interventions: Drug: ACP-196 (acalabrutinib)

INTERVENTIONS:
Drug: ACP-196 (acalabrutinib)

SUMMARY:
The purpose of this study is to characterize the safety and efficacy profile of ACP-196 (acalabrutinib) in subjects with relapsed or refractory Mantle Cell Lymphoma (MCL).

DETAILED DESCRIPTION:
This clinical trial is a Phase 2, multicenter, (approximately 70 global centers), open-label study in subjects with histologically documented MCL, who have relapsed after, or were refractory to, ≥ 1 (but not > 5) prior treatment regimens. Subjects will be enrolled and will take 100 mg of acalabrutinib twice per day (BID) in repeated 28-day cycles.

Treatment with acalabrutinib may be continued until disease progression or an unacceptable drug-related toxicity occurs. Dose modification provisions are provided in the study protocol.

All subjects will have hematology, chemistry, and urinalysis safety panels done at screening. Once dosing commences (Day 1), all subjects will be evaluated for safety, including serum chemistry and hematology, once weekly for the first 4 weeks, every 2 weeks in Cycle 2, every 4 weeks in Cycles 3 to 12, and every 24 weeks thereafter. PK/PD testing will be done in Cycles 1 and 2. Tumor assessments will be completed at 8- to 24-week intervals during the trial.

ELIGIBILITY:
Inclusion criteria:

* Men and women ≥ 18 years of age.
* Pathologically confirmed MCL, with documentation of monoclonal B cells that have a chromosome translocation t(11;14)(q13;q32) and/or overexpress cyclin D1.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
* Agreement to use contraception during the study and for 30 days after the last dose of study drugs if sexually active and able to bear or beget children.

Exclusion criteria:

* A life-threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ACP-196 (acalabrutinib), or put the study outcomes at undue risk
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification, or corrected QT interval (QTc) > 480 msec.
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.
* Breast feeding or pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2015-03-02 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2026-09-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Acerta Pharma, Study Director — 1-888-292-9613
Locations (56):
- United States (9):
  - Research Site, Tampa, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Niles, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Boston, Massachusetts
  - Research Site, Hackensack, New Jersey
  - Research Site, New York, New York
  - Research Site, Houston, Texas
  - Research Site, Seattle, Washington
- Australia (3):
  - Research Site, Monash
  - Research Site, Sydney
  - Research Site, Wodonga
- Belgium (4):
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Liège
  - Research Site, Yvoir
- Research Site, Prague, Czechia
- France (20):
  - Research Site, Angers
  - Research Site, Caen
  - Research Site, Clermond Ferrand
  - Research Site, Créteil
  - Research Site, Dijon
  - Research Site, Grenoble
  - Research Site, La Roche - Sure-Yon
  - Research Site, Lille
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Pierre-Bénite
  - Research Site, Rennes
  - Research Site, Rouen
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Strasbourg
  - Research Site, Toulouse
  - Research Site, Tours
  - Research Site, Vandœuvre-lès-Nancy
- Italy (4):
  - Research Site, Bologna
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Novara
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Maastricht
  - Research Site, Rotterdam
- Poland (3):
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Olsztyn
- Spain (2):
  - Research Site, Badalona
  - Research Site, Pamplona
- United Kingdom (7):
  - Research Site, Cardiff
  - Research Site, Leeds
  - Research Site, Leicester
  - Research Site, Nottingham
  - Research Site, Oxford
  - Research Site, Plymouth
  - Research Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Wang M, Rule S, Zinzani PL, Goy A, Casasnovas O, Smith SD, Damaj G, Doorduijn J, Lamy T, Morschhauser F, Panizo C, Shah B, Davies A, Eek R, Dupuis J, Jacobsen E, Kater AP, Le Gouill S, Oberic L, Robak T, Covey T, Dua R, Hamdy A, Huang X, Izumi R, Patel P, Rothbaum W, Slatter JG, Jurczak W. Acalabrutinib in relapsed or refractory mantle cell lymphoma (ACE-LY-004): a single-arm, multicentre, phase 2 trial. Lancet. 2018 Feb 17;391(10121):659-667. doi: 10.1016/S0140-6736(17)33108-2. Epub 2017 Dec 11. PMID 29241979
- See also: redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-LY-004&attachmentIdentifier=174abcea-afd1-4e70-80f7-35b2ebf5ffdb&fileName=ACE-LY-004_CSP-redacted.pdf&versionIdentifier=
- See also: redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-LY-004&attachmentIdentifier=d95872f9-fa74-4ce1-8ba3-a297d59adcc1&fileName=ACE-LY-004_CSR_Synopsis_redacted.pdf&versionIdentifier=
- See also: redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-LY-004&attachmentIdentifier=34251c79-b079-49d9-893d-ad2b1853f487&fileName=ACE-LY-004_SAP_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For the ACE-LY-004 program, Study Terminated by Sponsor refers to the following: Patients receiving treatment benefits will continue to be provided with study medication in the Post Final Analysis Management of the trial. No further data collection for analysis and reporting will be completed after the final Analysis.
Groups:
- ACP-196 100 mg BID: subjects with relapsed/refractory MCL
Period: Overall Study
Arm/Group | ACP-196 100 mg BID
Started | 124
Completed | 0
Not Completed | 124
Not completed — Death | 59
Not completed — Withdrawal by Subject | 10
Not completed — study terminated by sponsor | 51
Not completed — Lost to Follow-up | 3
Not completed — SITE CLOSURE - PI RETIREMENT | 1

BASELINE CHARACTERISTICS:
Population: The analysis population included All Treated Subjects.
Arm/Group | ACP-196 100 mg BID
Number analyzed (Participants) | 124
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.1 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 99
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 90
  Not Reported | 30
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Black or African American | 3
  Native Hawaiian or Other Pacific Islander | 0
  White | 92
  Not Reported | 29
Region of Enrollment [Number; unit: Participants]
  Australia | 2
  Belgium | 2
  France | 26
  Italy | 8
  Netherlands | 5
  Poland | 19
  Spain | 4
  United Kingdom | 13
  USA | 45

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) of ACP-196 (Acalabrutinib) in Subjects With Previously Treated MCL.
Description: The overall response rate (ORR) is defined as the proportion of subjects achieving either a partial remission (response) (PR) or complete response (CR) according to the Lugano Classification for NHL (Cheson 2014) as assessed by investigators, where SD stands for Stable Disease, PD for Progressive Disease and NE for Not Evaluable.
Time Frame: From the date of the first dose until 30 days after the last dose of the study drug or start of a new anti-cancer treatment, whichever came first, assessed up to approximately 4 year and 10 months. 1 cycle =28 days
Population: The analysis population included all treated subjects.
Measure: Count of Participants; unit: Participants
Groups:
- ACP-196 (Acalabrutinib): ACP-196 (acalabrutinib) 100 mg BID
Arm/Group | ACP-196 (Acalabrutinib)
Number analyzed (Participants) | 124
Participants
  CR | 59
  PR | 42
  SD | 10
  PD | 10
  NE | 3

ADVERSE EVENTS:
Time Frame: From the date of the first dose until 30 days after the last dose of the study drug or start of a new anti-cancer treatment, whichever came first, assessed up to approximately 4 year and 10 months.
Groups:
- ACP-196 100 mg BID: Description (Arm-group)
Arm/Group | ACP-196 100 mg BID
All-Cause Mortality (participants affected / at risk) | 59/124
Serious Adverse Events (participants affected / at risk) | 62/124
Other Adverse Events (participants affected / at risk) | 122/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACP-196 100 mg BID (N=124)
Anaemia (Blood and lymphatic system disorders) | 6 (9)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Leukostasis syndrome (Blood and lymphatic system disorders) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chest pain (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 4 (4)
Non-cardiac chest pain (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Jaundice extrahepatic obstructive (Hepatobiliary disorders) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (2)
Escherichia infection (Infections and infestations) | 1 (2)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (1)
Paronychia (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 8 (8)
Pseudomonal bacteraemia (Infections and infestations) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Streptococcal bacteraemia (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (2)
Urinary tract infection bacterial (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1)
General physical condition abnormal (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Autoimmune encephalopathy (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (2)
Suicide attempt (Psychiatric disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (2)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACP-196 100 mg BID (N=124)
Anaemia (Blood and lymphatic system disorders) | 16 (25)
Haemolysis (Blood and lymphatic system disorders) | 1 (1)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1 (1)
Increased tendency to bruise (Blood and lymphatic system disorders) | 3 (3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 14 (18)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (11)
Angina pectoris (Cardiac disorders) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1)
Right ventricular enlargement (Cardiac disorders) | 1 (1)
Sinus arrest (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 2 (2)
Otorrhoea (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 4 (4)
Vertigo positional (Ear and labyrinth disorders) | 2 (3)
Hyperparathyroidism (Endocrine disorders) | 1 (1)
Cataract (Eye disorders) | 4 (5)
Chalazion (Eye disorders) | 1 (2)
Conjunctival haemorrhage (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 5 (7)
Eye discharge (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1)
Eyelid rash (Eye disorders) | 1 (1)
Lacrimation increased (Eye disorders) | 7 (13)
Ocular hyperaemia (Eye disorders) | 1 (1)
Periorbital swelling (Eye disorders) | 1 (1)
Scleral hyperaemia (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 8 (11)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 14 (21)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 10 (11)
Aerophagia (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 20 (26)
Dental caries (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 47 (76)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 3 (3)
Food poisoning (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal mucosa hyperaemia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal polyp (Gastrointestinal disorders) | 1 (1)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (8)
Glossodynia (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Hyperchlorhydria (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 3 (3)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 27 (49)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Oesophageal spasm (Gastrointestinal disorders) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 2 (4)
Proctalgia (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 9 (17)
Tooth disorder (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 18 (30)
Asthenia (General disorders) | 22 (35)
Chest discomfort (General disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Chills (General disorders) | 4 (4)
Crepitations (General disorders) | 1 (1)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 37 (70)
Gait disturbance (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 3 (3)
Influenza like illness (General disorders) | 6 (10)
Malaise (General disorders) | 1 (1)
Nodule (General disorders) | 2 (3)
Non-cardiac chest pain (General disorders) | 4 (4)
Oedema (General disorders) | 2 (2)
Oedema peripheral (General disorders) | 11 (16)
Pain (General disorders) | 4 (4)
Peripheral swelling (General disorders) | 7 (8)
Pyrexia (General disorders) | 19 (26)
Sensation of foreign body (General disorders) | 1 (1)
Suprapubic pain (General disorders) | 1 (1)
Swelling (General disorders) | 2 (2)
Vessel puncture site haematoma (General disorders) | 1 (2)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1)
Contrast media allergy (Immune system disorders) | 1 (1)
Food allergy (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (2)
Hypogammaglobulinaemia (Immune system disorders) | 2 (2)
Seasonal allergy (Immune system disorders) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 11 (12)
Bronchitis viral (Infections and infestations) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2)
Chronic sinusitis (Infections and infestations) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Conjunctivitis (Infections and infestations) | 4 (4)
Cystitis (Infections and infestations) | 1 (1)
Cytomegalovirus viraemia (Infections and infestations) | 1 (1)
Dacryocystitis (Infections and infestations) | 1 (1)
Dermatitis infected (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1)
Eye infection (Infections and infestations) | 2 (2)
Fungal infection (Infections and infestations) | 2 (2)
Fungal skin infection (Infections and infestations) | 1 (2)
Furuncle (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 1 (1)
Herpes dermatitis (Infections and infestations) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 10 (10)
Infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 7 (7)
Jc virus infection (Infections and infestations) | 1 (1)
Laryngitis (Infections and infestations) | 4 (5)
Localised infection (Infections and infestations) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 6 (13)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (1)
Mastoiditis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 10 (14)
Ophthalmic herpes zoster (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 3 (3)
Otitis externa (Infections and infestations) | 1 (1)
Otosalpingitis (Infections and infestations) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 1 (1)
Peripheral nerve infection (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 8 (9)
Pulpitis dental (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 3 (3)
Rhinitis (Infections and infestations) | 6 (6)
Rhinovirus infection (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 16 (25)
Skin infection (Infections and infestations) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Tracheitis (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 20 (30)
Urinary tract infection (Infections and infestations) | 5 (13)
Vascular device infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 16 (23)
Fall (Injury, poisoning and procedural complications) | 6 (6)
Hand fracture (Injury, poisoning and procedural complications) | 1 (2)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (3)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1)
Vaccination complication (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2)
Blood cholesterol increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 3 (5)
Blood iron decreased (Investigations) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Blood urea increased (Investigations) | 1 (1)
Breath sounds abnormal (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 4 (5)
Platelet count decreased (Investigations) | 3 (3)
Serum ferritin decreased (Investigations) | 1 (1)
Thyroxine decreased (Investigations) | 1 (1)
Transaminases increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 4 (6)
Weight increased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 8 (12)
Dehydration (Metabolism and nutrition disorders) | 3 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (6)
Hyperuricaemia (Metabolism and nutrition disorders) | 5 (6)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (8)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (2)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (16)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (15)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Groin pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 (3)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 (12)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 (11)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 27 (49)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (9)
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (6)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3)
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1)
Balance disorder (Nervous system disorders) | 2 (2)
Burning sensation (Nervous system disorders) | 2 (2)
Carotid arteriosclerosis (Nervous system disorders) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Disturbance in attention (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 18 (21)
Dizziness postural (Nervous system disorders) | 1 (3)
Dysgeusia (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 48 (60)
Hypoaesthesia (Nervous system disorders) | 7 (9)
Intention tremor (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 9 (12)
Migraine (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 3 (4)
Neuropathy peripheral (Nervous system disorders) | 2 (2)
Paraesthesia (Nervous system disorders) | 10 (11)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Presyncope (Nervous system disorders) | 3 (3)
Resting tremor (Nervous system disorders) | 1 (2)
Sciatica (Nervous system disorders) | 4 (4)
Sensory loss (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 5 (5)
Tremor (Nervous system disorders) | 2 (2)
Device occlusion (Product Issues) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 9 (9)
Mental status changes (Psychiatric disorders) | 1 (1)
Sleep disorder (Psychiatric disorders) | 4 (4)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (4)
Pollakiuria (Renal and urinary disorders) | 4 (4)
Renal failure (Renal and urinary disorders) | 2 (2)
Renal injury (Renal and urinary disorders) | 1 (1)
Strangury (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (3)
Urinary retention (Renal and urinary disorders) | 2 (2)
Adnexa uteri pain (Reproductive system and breast disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 2 (2)
Prostatitis (Reproductive system and breast disorders) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 29 (38)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 (26)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Middle lobe syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 (10)
Pulmonary air leakage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Blood blister (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 4 (5)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 7 (7)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 1 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 11 (14)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6)
Purpura (Skin and subcutaneous tissue disorders) | 6 (7)
Rash (Skin and subcutaneous tissue disorders) | 18 (31)
Rash erythematous (Skin and subcutaneous tissue disorders) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 (3)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 3 (4)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Aortic stenosis (Vascular disorders) | 1 (1)
Arterial disorder (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 8 (8)
Hot flush (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 4 (5)
Hypotension (Vascular disorders) | 6 (6)
Lymphoedema (Vascular disorders) | 2 (2)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 1 (1)
Peripheral venous disease (Vascular disorders) | 1 (2)
Thrombophlebitis superficial (Vascular disorders) | 1 (1)
Thrombosed varicose vein (Vascular disorders) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/26/NCT02213926/Prot_002.pdf
  • Statistical Analysis Plan (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/26/NCT02213926/SAP_003.pdf